CLINICAL TRIAL: NCT05867290
Title: Mindful Music-listening to as a Tool to Improve Sleep Post-stroke: A Single Case Experimental Design Study
Brief Title: Music for Sleep After Stroke
Acronym: MUSAS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other); University of Edinburgh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GN22ST470
Record Dates: First submitted 2023-02-16; First posted 2023-05-19 (Actual); Last update posted 2023-05-19 (Actual); Status verified 2023-05

CONDITIONS: Stroke; Cardiovascular Diseases; Brain Diseases; Vascular Diseases; Insomnia; Sleep Disorder; Sleep Disturbance
MeSH Terms: conditions — Stroke; Cardiovascular Diseases; Brain Diseases; Vascular Diseases; Sleep Initiation and Maintenance Disorders; Sleep Wake Disorders; Parasomnias

STUDY DESIGN:
Intervention Model Description: Single Case Experimental Design (SCED) methodology using multiple baseline across participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Baseline Phase (No Intervention): Randomly allocated baseline phase (no intervention) of 7, 11 or 15 days.
- Intervention Phase (Experimental): 5 week mindful-music listening intervention including sleep hygiene
  Interventions: Behavioral: Mindful music-listening with sleep hygiene

INTERVENTIONS:
Behavioral: Mindful music-listening with sleep hygiene — 5 week intervention consisting of sleep hygiene (week 1) and daily bedtime mindful music-listening for 30 minutes or until about to fall asleep, if sooner (weeks 2-5)
  Arms: Intervention Phase

SUMMARY:
Sleep difficulties are common following stroke yet effective evidence-based interventions for improving sleep in this population are lacking. A small number of studies have investigated the use of music listening as a way to improve sleep in adults with insomnia.

This study aims to examine whether a mindful music-listening intervention can reduce subjective and objective insomnia symptoms and improve mood and fatigue post-stroke.

Six adults with a clinical diagnosis of stroke presenting with an insomnia disorder will be recruited from stroke services within NHS Greater Glasgow and Clyde. A multiple baseline single case experimental design will be employed. Participants will be randomly allocated to a baseline phase of 7, 11 or 15 days, followed by a five-week mindful music-listening intervention incorporating sleep hygiene. Changes in subjective and objective sleep will be measured using questionnaires and actigraphy, respectively. Mood and fatigue will also be measured. The data will be analysed using visual inspection, Tau-U and multi-level modelling.

ELIGIBILITY:
Inclusion Criteria:

* aged 18+ (no upper age limit);
* clinically and/or radiologically confirmed diagnosis of stroke
* score of ≤16 on the Sleep Condition Indicator (SCI; (Espie et al, 2018))
* at least 3-months post-stroke

Exclusion Criteria:

* Transient Ischemic Attack
* subarachnoid hemorrhage
* sleep medication commenced within the last 2 weeks (stable medication accepted)
* significant receptive aphasia or major psychiatric/substance abuse problem preventing engagement in the intervention
* deafness or severe hearing impairment preventing engagement in the intervention (use of hearing aids does not lead to exclusion where these support sufficient level of hearing for engagement)
* unable to give informed consent.
* participation in another intervention study with risk of contamination of study outcomes (determined on a case-by-case basis)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Sleep onset latency (SOL) | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Time taken to fall asleep in minutes measured using actigraphy and a sleep diary completed by the participant. Higher scores indicate greater SOL.

SECONDARY OUTCOMES:
Total sleep time (TST) | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Total time spent asleep in bed in minutes. Measured using actigraphy and a sleep diary completed by the participant. Higher scores indicated longer time spent asleep.
Wake after sleep onset (WASO) | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Total time spent awake after sleep onset in minutes. Measured using actigraphy and a sleep diary completed by the participant. Higher scores indicate longer time spent awake.
Number of night time awakenings | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Total number of awakenings during the night. Measured using actigraphy and a sleep diary completed by the participant. Min = 0 - no Max. Lower scores indicate fewer night time awakenings.
Time in bed (TIB) | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Total time spent in bed in minutes with higher scores indicating longer time spent in bed. Measured using a sleep diary completed by the participant.
Sleep restoration | Measured daily, from baseline to follow-up (day 1 up to day day 71).
  Participant rated level of sleep restoration on awakening. Measured using a 3-point scale: refreshed, somewhat refreshed, fatigued.
Insomnia classification | Completed at baseline, end of intervention (week 1 to weeks 6-8 and at follow up (3 weeks post-intervention)
  Sleep Condition Indicator (SCI) score. Min score= 0 - Max= 32 with lower scores indicating poorer sleep.
Daytime sleepiness | Completed at baseline, at the end of intervention (week 1 to weeks 6-8) and at follow-up (3 weeks post-intervention)
  Epworth Sleepiness Scale (ESS) score. Min score= 0 - Max= 24 with higher scores indicating greater levels of daytime sleepiness.
Anxiety symptoms | Completed at baseline, end of intervention (week 1 to weeks 6-8 and at follow up (3 weeks post-intervention)
  Generalized Anxiety Disorder Questionnaire (GAD-7) score. Min= 0 - Max= 21 with higher scores indicating more severe symptoms.
Depressive symptoms | Completed at baseline, end of intervention (week 1 to weeks 6-8 and at follow up (3 weeks post-intervention)
  Patient Health Questionnaire (PhQ-9) score. Min= 0 - Max= 27 with higher scores indicating more severe symptoms.
Fatigue | Completed at baseline, end of intervention (week 1 to weeks 6-8 and at follow up (3 weeks post-intervention)
  Fatigue Severity Scale (FSS) score. Min= 9 - Max= 63 with higher scores indicating greater fatigue severity.
Adherence | Completed daily by the participant during the intervention music listening phase (weeks 3-5 to weeks 8-10)
  Adherence to mindful music-listening as measured through music listening diary. Min= 0 - Max= 28 with higher scores indicating greater adherence.

CONTACTS AND LOCATIONS:
Locations (1):
- Greater Glasgow and Clyde Stroke Services, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: No